CLINICAL TRIAL: NCT01813396
Title: Prediction of Functional Disability and Randomized Clinical Trial in Subjects With Stiff Shoulders: Joint Mobility, Range of Motion, Muscle Stiffness, and Shoulder Physical Activity
Brief Title: Prediction of Functional Disability and Clinical Trial in Subjects With Stiff Shoulders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201012075RB
Record Dates: First submitted 2013-02-20; First posted 2013-03-19 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Muscle Stiffness
Keywords: shoulder; muscle stiffness; shoulder physical activity; range of motion; joint mobility
MeSH Terms: interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- joint mobilization/massage (Experimental): joint mobilization: End-range joint mobilization
  massage: massage twice a week on the identified muscle(s) of the involved shoulder about 6 minutes for each muscle for 3 months. The techniques of massage include petrissage for 3 minutes and rolling for 3 minutes of soft tissues
  Interventions: Other: joint mobilization plus massage
- joint mobilization/shoulder physical activity guide (Experimental): joint mobilization: End-range joint mobilization shoulder physical activity guide: shoulder physical activity guide is based on the appropriate cut off activity level identified in the predication rule
  Interventions: Other: joint mobilization/shoulder physical activity guide

INTERVENTIONS:
Other: joint mobilization plus massage
  Arms: joint mobilization/massage
Other: joint mobilization/shoulder physical activity guide
  Arms: joint mobilization/shoulder physical activity guide

SUMMARY:
First, the purpose of the first year study will examine the joint capsule/muscular and shoulder physical activity hypotheses related to ROM deficits as well as functional disability in subjects with Stiff shoulders. Second, the purpose of the second and third year study will investigate the long-term effect of 12-week joint mobilization, 12-week joint mobilization plus soft tissue mobilization/massage, and 12-week joint mobilization plus soft tissue mobilization/massage with appropriate shoulder physical activity guide on subjects with Stiff shoulders. Subjects: First year: thirty subjects with Stiff shoulders will be recruited. Second and third years: forty-five subjects with Stiff shoulders for one year follow-up. Methods: For the measurement outcomes; functional disability, rotation range of motion, joint mobility, muscle stiffness, and shoulder physical activity will be measured by self-reported Flexi-level Scale of Shoulder Function or performance-based motion analysis, goniometer, uni-axis load cell and electromagnetic tracking sensor, myotonometer, and accelerometers, respectively.

ELIGIBILITY:
Inclusion Criteria:

* [1] a limited ROM of flexion, abduction, and rotation (ROM < 20% to the sound side); and [2] pain and stiffness in the shoulder region for at least 3 months.

Exclusion Criteria:

* surgery on the particular shoulder, [2] rheumatoid arthritis, [3] stroke with residual shoulder involvement, [4] fracture of the shoulder complex, [5] rotator cuff deficiency, and [6] resting pain, intolerable pain, or muscle spasm during active and/or passive motion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
shoulder physical activity | right after 12-week treatment
  analysis by RT3(shoulder activity measurement device)

SECONDARY OUTCOMES:
Muscle stiffness | right after 12-week treatment
  analysis by myotonometer(muscle stiffness measurement device)

OTHER OUTCOMES:
Joint play assessment | right after 12-week treatment
  joint play scale measured by physical therapist

CONTACTS AND LOCATIONS:
Overall Officials: jiu-jenq Lin, PhD, Principal Investigator — Natinal Taiwan University Hospital
Locations (1):
- Physical Therapy Center or Department of Physical Medicine and Rehabilitation at National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Yang JL, Lin JJ, Huang HY, Huang TS, Chao YW. Shoulder physical activity, functional disability and task difficulties in patients with stiff shoulders: interpretation from RT3 accelerator. Man Ther. 2014 Aug;19(4):349-54. doi: 10.1016/j.math.2014.02.005. Epub 2014 Mar 5. PMID 24650638